CLINICAL TRIAL: NCT01489293
Title: Characterization of the Expression and Activity of Inhibitory Receptors Such as CLM-1 in Eosinophils of Atopic Subjects
Brief Title: Inhibitory Receptors in Eosinophils of Atopic Subjects
Status: Completed | Type: Observational
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: MMC110053CTIL
Record Dates: First submitted 2011-12-07; First posted 2011-12-09 (Estimated); Last update posted 2018-03-22 (Actual); Status verified 2018-03

CONDITIONS: Atopy; Atopic Dermatitis; Asthma; Allergic Rhinitis; Food Allergy
MeSH Terms: conditions — Dermatitis, Atopic; Asthma; Rhinitis, Allergic; Food Hypersensitivity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- atopic subjects: Patients with one atopic disease or more (atopic dermatitis,rhinitis, asthma, food allergy)
- non-atopic subjects: Control group without atopic diseases.

SUMMARY:
The purpose of this study is to analyze the expression and activity of inhibitory molecules on eosinophils obtained from allergic subjects.

ELIGIBILITY:
Inclusion Criteria:

* age 20-60 years
* a physician-diagnosed atopic disease

Exclusion Criteria:

* atopic disease not active
* steroid treatment
* active non-atopic inflammatory disease, including infections
* pregnancy

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: allergy clinic
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2012-05-01 (Actual); Primary Completion 2013-12-31 (Actual); Study Completion 2013-12-31 (Actual)

PRIMARY OUTCOMES:
Expression of surface molecules on eosinophils as assessed by flow cytometry | December 2013
  Blood samples from donors will be stained and evaluated by flow cytomtery

CONTACTS AND LOCATIONS:
Overall Officials: Alon Y Hershko, MD, PhD, Principal Investigator — Meir Medical Center
Locations (1):
- Meir Medical Center. Unit of Allergy and Clinical Immunology, Kfar Saba, Israel